CLINICAL TRIAL: NCT07184684
Title: Sinonasal Microbiome Transplant as a Therapy for Chronic Rhinosinusitis (CRS): A Randomized , Placebo Controlled Cross Over Trial
Brief Title: Sinonasal Microbiome Transplant as a Therapy for Chronic Rhinosinusitis (CRS).
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2024-03308-02
Record Dates: First submitted 2024-07-12; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps; Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Intervention Model Description: All participants will run through the study twice with a 7 month wash-out in between. Once the participant will run through the microbiome translant arm and once through the placebo arm.. Participants and investigators will be blinded to the if the participant gets microbiome transplantation or placebo.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiome transplant (Active Comparator): The study subject is examined before and after recieving 13 days of antibiotics followed by 5 concecutive days of microbiome transplant.
  Interventions: Procedure: Sinonasal microbiome transplant procedure.
- Placebo transplant (Placebo Comparator): The study subject is examined before and after recieving 13 days of antibiotics followed by 5 concecutive days of placebo (saline) transplant.
  Interventions: Other: Placebo saline transplant

INTERVENTIONS:
Procedure: Sinonasal microbiome transplant procedure. — A sinonasal microbiome transplant obtained from a healthy donor and administered as a nasal lavage once daily for five consecutive days.
  Arms: Microbiome transplant
Other: Placebo saline transplant — Placebo transplant containing saline administered as a nasala lavage once daily for five consecutive days.
  Arms: Placebo transplant

SUMMARY:
Chronic rhinosinusitis (CRS) is a disease associated with impaired quality of life and substantial societal costs. Much is still uncertain regarding the underlying etiology of the disease. Current treatment protocols are based on observed effects rather than a mechanistic understanding of the disease and thus patients often report unsatisfactory symptom reduction despite treatment with maximal medical therapy and even surgery.

CRS is subgrouped phenotypically based on whether or not polyps are observed. Recently an endotypical differentiation reflecting the underlying inflammatory profile has been recommended as well, especially for research.

Increasing interest in the role of the commensal microbiome inflammatory diseases has followed a growing understanding of its profound impact on the human immune system. Current research indicates that instability and dysfunction of the microbiome is linked to inflammatory disease rather than compositional differences. Previous research has shown that microbiome transplants are effective in restoring the commensal microbiome and reducing inflammation in gastrointestinal disease and in a previous pilot study the investigators showed that sinonasal microbiome transplants are feasible and were associated with reduced symptoms in chronic rhinosinusitis without nasal polyps (CRSsNP).

This study will examine if the positive effect on patients symptoms observed in a previous pilot study are sustained in a placebo controlled, blinded study. In addition to this the study will also examine any differences in microbiome structure, stability, and function between patients with CRS and healthy donors as well as any correlation to disease phenotype or inflammatory endotype.

ELIGIBILITY:
Inclusion Criteria (CRS-Patients):

* 2 nasal symptoms, 1 of which must be nasal obstruction or discolored discharge.
* Sinusitis verified by endoscopy or CT scan
* Duration > 12 weeks.
* Signed informed consent to participate in the study.

Exclusion Criteria (CRS-Patients):

* Antibiotic treatment in the last 3 months before study start.
* Ongoing or recent participation in another clinical trial.
* Any medication that might affect the results in an unpredictable manner.
* Treatment with monoclonal antibodies (biologics).
* Immunodeficiency other than low grade MBL deficiency.
* Pregnancy or breastfeeding
* Severe anatomical abnormalities.
* SNOT 22 < 20.

Inclusion Criteria (Donors):

* No history of sinonasal or lower airway disease within the last two years other than the common cold.
* Accepted as a donor by the patient.
* Signed informed consent to participate in the study.

Exclusion Criteria (CRS-Patients):

* Chronic rhinosinusitis.
* Acute rhinosinusitis within the last two years.
* Nasal polyposis
* Antibiotic treatment within the last 3 months before the study start.
* On going or recent participation in another clinical trial.
* Findings in the pre study scan that makes the donor unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Sino-nasal outcome test 22 (SNOT-22) (min 0 - max 110 higher being worse) | 14 days before intervention, on the first day of intervention, 2 and 3 months after intervention and as a follow up 1, 2 and 3 years after the study.
  Subjective symptom grading of the patients will be used to asses efficacy of the treatment and the duration of the treatment effect.

SECONDARY OUTCOMES:
Endoscopy | 2 weeks before intervention, 3 months after intervention and as a follow up 1, 2 and 3 years after the study.
  Patients will be documented using video endoscopy for later, blinded grading.
Total Nasal Symptom Score. (min 0 - max 9) | 14 days before intervention, daily during the five days of intervention, 2 and 3 months after intervention and as a follow up 1, 2 and 3 years after the study.
  The TNSS scale will be used to measure nasal symptoms of donors and patients especially during the transplant procedure to evaluate the tolerability of the procedure.
Metagenomics | 6 and 2 weeks before intervention, 8 and 12 weeks after intervention and as a follow up twice with 4 weeks apart 1, 2 and 3 years after the study.
  Microbiological samples will be collected from both donors and patients to assess whether the microbiota differ in patients with CRS compared to healthy subjects regarding composition, abundance, diversity, and stability. Further we will examine the effect of the microbiome transplant procedure on the recipients microbiota.
Metabolomics | 2 weeks before intervention and 12 weeks after intervention and as a follow up 1, 2 and 3 years after the study.
  Metabolomics samples will be collected from both donors and patients to assess if the microbiome activity differ in patients with CRS compared to healthy subjects and if this activity is affected by the microbiome transplant procedure.
Inflammatory markers | 2 weeks before intervention, 12 weeks after intervention and as a follow up 1, 2 and 3 years after the study.
  Biopsies from the nasal mucosa will be collected from both donors and patients and analysed for inflammatory endotypes and to assess the effect of the microbiome transplant procedure in the patients.
Adverse events | Entire study duration. Total study duration is 1 year and 5 months for the study and 3 years of follow up.
  Any adverse events reported by the patients will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Mårtensson, MD, PhD, Principal Investigator — Region Skåne, Lund University
Locations (1):
- Departement of ORL, Helsingborg, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will be presented on group level.

REFERENCES:
- [Background] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Background] Rudmik L, Smith TL. Quality of life in patients with chronic rhinosinusitis. Curr Allergy Asthma Rep. 2011 Jun;11(3):247-52. doi: 10.1007/s11882-010-0175-2. PMID 21234819
- [Background] Wahid NW, Smith R, Clark A, Salam M, Philpott CM. The socioeconomic cost of chronic rhinosinusitis study. Rhinology. 2020 Apr 1;58(2):112-125. doi: 10.4193/Rhin19.424. PMID 32172284
- [Background] McCormick JP, Thompson HM, Cho DY, Woodworth BA, Grayson JW. Phenotypes in Chronic Rhinosinusitis. Curr Allergy Asthma Rep. 2020 May 19;20(7):20. doi: 10.1007/s11882-020-00916-6. PMID 32430653
- [Background] Kato A, Peters AT, Stevens WW, Schleimer RP, Tan BK, Kern RC. Endotypes of chronic rhinosinusitis: Relationships to disease phenotypes, pathogenesis, clinical findings, and treatment approaches. Allergy. 2022 Mar;77(3):812-826. doi: 10.1111/all.15074. Epub 2021 Sep 15. PMID 34473358
- [Background] Stevens WW, Peters AT, Tan BK, Klingler AI, Poposki JA, Hulse KE, Grammer LC, Welch KC, Smith SS, Conley DB, Kern RC, Schleimer RP, Kato A. Associations Between Inflammatory Endotypes and Clinical Presentations in Chronic Rhinosinusitis. J Allergy Clin Immunol Pract. 2019 Nov-Dec;7(8):2812-2820.e3. doi: 10.1016/j.jaip.2019.05.009. Epub 2019 May 22. PMID 31128376
- [Background] Foster KR, Schluter J, Coyte KZ, Rakoff-Nahoum S. The evolution of the host microbiome as an ecosystem on a leash. Nature. 2017 Aug 2;548(7665):43-51. doi: 10.1038/nature23292. PMID 28770836
- [Background] Belkaid Y, Hand TW. Role of the microbiota in immunity and inflammation. Cell. 2014 Mar 27;157(1):121-41. doi: 10.1016/j.cell.2014.03.011. PMID 24679531
- [Background] Martens K, Pugin B, De Boeck I, Spacova I, Steelant B, Seys SF, Lebeer S, Hellings PW. Probiotics for the airways: Potential to improve epithelial and immune homeostasis. Allergy. 2018 Oct;73(10):1954-1963. doi: 10.1111/all.13495. Epub 2018 Jun 28. PMID 29869783
- [Background] Aggarwal N, Kitano S, Puah GRY, Kittelmann S, Hwang IY, Chang MW. Microbiome and Human Health: Current Understanding, Engineering, and Enabling Technologies. Chem Rev. 2023 Jan 11;123(1):31-72. doi: 10.1021/acs.chemrev.2c00431. Epub 2022 Nov 1. PMID 36317983
- [Background] Psaltis AJ, Mackenzie BW, Cope EK, Ramakrishnan VR. Unraveling the role of the microbiome in chronic rhinosinusitis. J Allergy Clin Immunol. 2022 May;149(5):1513-1521. doi: 10.1016/j.jaci.2022.02.022. Epub 2022 Mar 14. PMID 35300985
- [Background] Paramasivan S, Bassiouni A, Shiffer A, Dillon MR, Cope EK, Cooksley C, Ramezanpour M, Moraitis S, Ali MJ, Bleier B, Callejas C, Cornet ME, Douglas RG, Dutra D, Georgalas C, Harvey RJ, Hwang PH, Luong AU, Schlosser RJ, Tantilipikorn P, Tewfik MA, Vreugde S, Wormald PJ, Caporaso JG, Psaltis AJ. The international sinonasal microbiome study: A multicentre, multinational characterization of sinonasal bacterial ecology. Allergy. 2020 Aug;75(8):2037-2049. doi: 10.1111/all.14276. Epub 2020 Mar 30. PMID 32167574
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Wang ZK, Yang YS, Chen Y, Yuan J, Sun G, Peng LH. Intestinal microbiota pathogenesis and fecal microbiota transplantation for inflammatory bowel disease. World J Gastroenterol. 2014 Oct 28;20(40):14805-20. doi: 10.3748/wjg.v20.i40.14805. PMID 25356041
- [Background] Martensson A, Cervin-Hoberg C, Huygens F, Lindstedt M, Sakellariou C, Greiff L, Cervin A. Upper airway microbiome transplantation for patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2023 Jun;13(6):979-988. doi: 10.1002/alr.23122. Epub 2023 Jan 1. PMID 36515012
- [Background] Martensson A, Abolhalaj M, Lindstedt M, Martensson A, Olofsson TC, Vasquez A, Greiff L, Cervin A. Clinical efficacy of a topical lactic acid bacterial microbiome in chronic rhinosinusitis: A randomized controlled trial. Laryngoscope Investig Otolaryngol. 2017 Nov 8;2(6):410-416. doi: 10.1002/lio2.93. eCollection 2017 Dec. PMID 29299516